CLINICAL TRIAL: NCT00132041
Title: Multicenter Feasibility Study of Percutaneous Radiofrequency Ablation of Hepatocellular Carcinoma in Cirrhotic Patients
Brief Title: Radiofrequency Ablation in Treating Patients With Liver Cancer and Cirrhosis
Acronym: ACRIN-6673
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American College of Radiology Imaging Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000439446; ACRIN-6673 (Other: CIP); U01CA080098 (NIH); U01CA079778 (NIH); NCT00399958 (obsolete NCT alias)
Record Dates: First submitted 2005-08-16; First posted 2005-08-19 (Estimated); Results first posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-08

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; localized unresectable adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- All Patients (Other): patients with cirrhosis undergoing solitary or repetitive percutaneous RFA treatment sessions for the treatment of HCC.
  Interventions: Device: radiofrequency ablation

INTERVENTIONS:
Device: radiofrequency ablation
  Other Names: RFA

SUMMARY:
RATIONALE: Radiofrequency ablation uses a high-frequency, electric current to kill tumor cells. CT-, MRI-, or ultrasound-guided radiofrequency ablation may be an effective treatment for liver cancer and cirrhosis.

PURPOSE: This phase II trial is studying how well radiofrequency ablation works in treating patients with liver cancer and cirrhosis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 18-month successful disease control rate, defined as no identifiable liver tumor by CT scan, in patients with hepatocellular carcinoma and cirrhosis treated with solitary or repetitive percutaneous radiofrequency ablation (RFA).

Secondary

* Correlate tumor size, MELD score, and the number of RFA treatments (solitary or repetitive) with the 18-month successful disease control rate in patients treated with this procedure.
* Determine the local and remote intrahepatic and extrahepatic tumor recurrence rates in patients treated with this procedure.
* Correlate local and remote intrahepatic and extrahepatic tumor recurrence rates with the 18-month successful disease control rate in patients treated with this procedure.
* Correlate tumor size with the local disease control rate in patients treated with this procedure.
* Correlate solitary or repetitive RFA with or without local/regional tumor control with the development of extrahepatic tumor in these patients.
* Determine the local tumor eradication rate, as determined by examination of whole liver specimens or CT scan, in patients treated with this procedure.

OUTLINE: This is a multicenter study. Patients are stratified according to hepatic dysfunction using the MELD score (< 15 vs 15-25 vs > 25).

Patients undergo placement of an ablation electrode percutaneously into the tumor(s) by CT scan, MRI, or ultrasound guidance. Patients then undergo percutaneous radiofrequency ablation (RFA) directly to the tumor(s) for 12 minutes. Patients undergo CT scan of the liver within 1 week after RFA treatment and then every 3 months for up to 18 months. Patients with residual or recurrent intrahepatic tumor(s) detectable on the 3-month or subsequent CT scan undergo repeat RFA as is technically feasible and clinically indicated for up to 15 months after initial RFA treatment.

After completion of study treatment, patients are followed at 1 day, 1 week, 1 month, and then every 3 months for up to 18 months.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of hepatocellular carcinoma (HCC), meeting 1 of the following criteria:

  * Histologically confirmed HCC
  * Discrete non-biopsied hepatic tumors, meeting 1 of the following criteria:

    * Hypervascular tumor > 2 cm by 2 imaging studies
    * Hypervascular tumor > 2 cm by a single imaging study AND alpha-fetoprotein ≥ 400 ng/mL
  * Discrete non-biopsied hypervascular hepatic tumors by 2 consecutive imaging studies (e.g., CT scan or MRI) with documented tumor growth > 1 cm in diameter
* Histologically confirmed cirrhosis OR typical findings of cirrhosis (i.e., nodular liver, splenomegaly, varices, or ascites) by CT scan and/or MRI scan
* Single hepatic tumor > 3.0 cm but ≤ 5.0 cm in diameter OR 3 or fewer hepatic tumors ≤ 3.0 cm in diameter

  * No excessive intrahepatic tumor burden (i.e., > 3 hepatic tumors OR a single hepatic tumor > 5 cm OR more than 3 vague hypervascular nodules > 1 cm)
* Tumor(s) ≥ 1 cm from the main, right, and left portal veins and hollow viscera

  * No hepatic or portal vein tumor invasion
* Tumor(s) > 1 cm treatable by percutaneous radiofrequency ablation
* No extrahepatic tumor
* Not a surgical candidate due to any of the following reasons:

  * Tumor in an unresectable location
  * Comorbid disease
  * Insufficient hepatic reserve

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* No uncorrectable coagulopathy

Hepatic

* Not specified

Renal

* Creatinine ≤ 2.0 mg/dL

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active symptomatic bacterial or fungal infection that is newly diagnosed and/or requires treatment
* No absolute contraindication to IV iodinated contrast (i.e., history of significant contrast reaction not mitigated by appropriate premedication)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior or concurrent chemotherapy for HCC
* No prior or concurrent chemoembolization for HCC

Endocrine therapy

* Not specified

Radiotherapy

* No prior or concurrent radiotherapy for HCC

Surgery

* No prior choledochoenteric anastomosis
* No prior sphincterotomy of duodenal papilla

Other

* No prior or concurrent cryoablation for HCC
* No other prior or concurrent therapy for HCC
* At least 7 days since prior aspirin
* At least 24 hours since prior ibuprofen
* At least 12 hours since prior low molecular weight heparin preparations

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-12; Primary Completion 2009-08 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald D. Dodd, MD, Study Chair — The University of Texas Health Science Center at San Antonio
Locations (18):
- United States (18):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Cancer Institute, Temple, Texas

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://clinicaltrials.gov/ct2/show/NCT00132041

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: patients with cirrhosis undergoing solitary or repetitive percutaneous radiofrequency ablation (RFA) treatment sessions for the treatment of HCC.
Period: Baseline
Arm/Group | All Patients
Started | 51
Eligible | 45
Completed | 45
Not Completed | 6
Not completed — Ineligible | 6
Period: 3 Months Post Ablation
Arm/Group | All Patients
Started | 45
Completed | 42
Not Completed | 3
Not completed — Transplant | 1
Not completed — Non-Protocol Treatment | 2
Period: 6 Months Post Ablation
Arm/Group | All Patients
Started | 42
Completed | 32
Not Completed | 10
Not completed — Withdrawal by Subject | 2
Not completed — Death | 2
Not completed — Transplant | 6
Period: 9 Months Post Ablation
Arm/Group | All Patients
Started | 32
Completed | 30
Not Completed | 2
Not completed — Death | 1
Not completed — Transplant | 1
Period: 12 Months Post Ablation
Arm/Group | All Patients
Started | 30
Completed | 26
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Not completed — Transplant | 1
Not completed — non-protocol Treatment | 1
Period: 15 Months Post Ablation
Arm/Group | All Patients
Started | 26
Completed | 18
Not Completed | 8
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Not completed — Transplant | 5
Not completed — Non-Protocol Treatment | 1
Period: 18 Months Post Ablation
Arm/Group | All Patients
Started | 18
Completed | 12
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Transplant | 1
Not completed — Non-Protocol Treatment | 3
Not completed — ExtraHepatic tumor | 1

BASELINE CHARACTERISTICS:
Population: Eligible patient with cirrhosis being treated with RFA for HCC
Arm/Group | All Patients
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 62 [40 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 31
  More than one race | 0
  Unknown or Not Reported | 7

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Successful Control of Disease at 18 Months
Description: Outcome is positive (success) if alive and no disease is observed by CT at 18 months post start of therapy Outcome is negative if the patient was deceased or disease was observed by CT at 18 months post start of therapy Success rate it the fraction of eligible patients who were alive and disease free at 18 months.
Time Frame: 18 months after start of therapy
Population: Patients not reaching 18mo were considered failures
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Eligible Patients: patients with cirrhosis undergoing solitary or repetitive percutaneous radiofrequency ablation (RFA) treatment sessions for the treatment of HCC.
Arm/Group | Eligible Patients
Number analyzed (Participants) | 45
proportion of participants | .18 [0.080 to 0.321]
Statistical Analysis 1: Comparison: Eligible Patients; logistic regression was used to estimate the success rate; Test type: Other; Success rate = 0.18, 95% CI 2-sided [0.091 to 0.317] — logistic regression model without correcting for the clustering effect
Statistical Analysis 2: Comparison: Eligible Patients; logistic regression model after specifying site as cluster (using GEE approach); Test type: Other; Success rate = 0.19, 95% CI 2-sided [0.136 to 0.252]

2. Secondary Outcome: Number of Participants With Success in Those Who Received Solitary vs Repetitive Radiofrequency Ablation
Description: this outcome measures the impact of Solitary vs repetitive radiofrequency ablation on success.
  Success is defined as the number of patients centrally determined to be alive and tumor-free 18 months after start of therapy, corrected for repetitive RFA.
Time Frame: 18 months after start of therapy
Population: of the 45 participants, 35 had single ablate therapy while 10 received multiple RFA sessions.
Measure: Count of Participants; unit: Participants
Groups:
- Solitary Ablation: patients with cirrhosis undergoing solitary percutaneous radiofrequency ablation (RFA) treatment sessions for the treatment of HCC.
- Repetitive Ablation: patients with cirrhosis undergoing repetitive percutaneous radiofrequency ablation (RFA) treatment sessions for the treatment of HCC.
Arm/Group | Solitary Ablation | Repetitive Ablation
Number analyzed (Participants) | 35 | 10
Participants
  Success | 5 | 3
  Failure | 30 | 7
Statistical Analysis 1: Comparison: Solitary Ablation; logistic regression was used to estimate the success rate; Test type: Other; Success rate = 0.18, 95% CI 2-sided [0.091 to 0.317] — logistic regression model without correcting for the clustering effect
Statistical Analysis 2: Comparison: Solitary Ablation; multivariate logistic regression model was fit using GEEs to correct for site clustering effects, in which, the response variable was success/failure at 18 months and the covariates were tumor size, whether or not a patient received repeated RFA, whether or not a local tumor recurrence occurred, whether or not a remote tumor occurrence occurred, and two common confounding factors - age and gender; Test type: Other; p = 0.0004, Generlaized estimating equations; Multivariate logistic model. P-value for number of RFA sessions dichotomized 1: more than 1; using the latter as the reference; Slope = -3.7913, 95% CI 2-sided [-5.9056 to -1.6769] — This estimate is for the effect of a single RFA sessions (v multiple sessions) in the multivariate model response:18 mo success/failure; covariates: tumor size,repeated RFA, local tumor recurrence, remote tumor occurrence, and age and gender

3. Secondary Outcome: Effect of Tumor Size on Successful Control of Disease at 18 Months
Description: Outcome is positive (success) if alive and no disease is observed by CT at 18 months post start of therapy Outcome is negative if the patient was deceased or disease was observed by CT at 18 months post start of therapy Success rate it the fraction of eligible patients who were alive and disease free at 18 months. Tumor size is a continuous variable as measured at imaging.
Time Frame: 18 months after start of therapy
Population: 8 participants has successful control at 18mo; 37 participants did not.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Eligible Patients
Number analyzed (Participants) | 45
centimeters
  Successful Control mean size: number analyzed (Participants) | 8
  Successful Control mean size | 2.80 (0.85)
  Failure mean size | 3.32 (1.26)
Statistical Analysis 1: Comparison: Eligible Patients; Effect of tumor size in the multivariate model with response:18 mo success/failure; covariates: tumor size,repeated RFA, local tumor recurrence, remote tumor occurrence, and age and gender; Test type: Other; p = 0.0221, Generlaized Estimating Equations; multivariate GEE model using logistic link; GEE = -0.9101, 95% CI 2-sided [-1.6894 to -0.1308] — Estimation parameter is for tumor size when controlling for other covariates

4. Secondary Outcome: Local Tumor Recurrence (Control) Rates
Description: local tumor control rate is defined as a tumor that was ablated and was not seen again within the 18 month period
Time Frame: 18 months after start of therapy
Measure: Number (95% Confidence Interval); unit: percentage recurring
Arm/Group | Eligible Patients
Number analyzed (Participants) | 45
percentage recurring | 0.51 [0.358 to 0.663]

5. Secondary Outcome: Impact of Tumor Size on Local Control Rates
Description: Lesion level local control is defined as a success if a tumor is ablated and does not recur in 18 mo.
Time Frame: 18 months after start of therapy
Population: local tumor control rate (No Recurrence) is defined as a tumor that was ablated and was not seen again
Measure: Mean (Standard Deviation); unit: cm
Units Other Than Participants: lesions
Arm/Group | Eligible Patients
Number analyzed (Participants) | 45
Number analyzed (lesions) | 60
cm
  No Recurrance: number analyzed (lesions) | 36
  No Recurrance | 2.4833 (0.999)
  Recurrance: number analyzed (lesions) | 24
  Recurrance | 2.9417 (0.8622)
Statistical Analysis 1: Comparison: Eligible Patients; the mean tumor size in the two groups, recurred and non recurred tumors, will be compared using a t-test assuming H0: recur=non-recurr; Test type: Other; p = 0.06, t-test, 2 sided — assuming unequal variance (Satterthwaite p); Mean Difference (Final Values) = -0.458, Standard Error of Mean 0.2496 — Difference represents the size of tumors that do no recur minus those that do

6. Secondary Outcome: Development of Extra-hepatic Tumor
Description: Whether or not extrahepatic tumors were seen at 18months post ablation will be compared with the number of RFA sessions.
Time Frame: 18 months after start of therapy
Measure: Count of Participants; unit: Participants
Groups:
- Extrahepatic Tumor: In this group, extrahepatic tumors were observed within 18 months of the initial ablation
- No Extrahepatic Tumors: In this group, no extrahepatic tumors were observed within 18 months of the initial RFA
Arm/Group | Extrahepatic Tumor | No Extrahepatic Tumors
Number analyzed (Participants) | 6 | 39
Participants
  1-RFA | 2 | 25
  Multiple RFA | 4 | 14

7. Secondary Outcome: Local Tumor Eradication Rate by Examination of Liver Via Autopsy or Transplant vs That Determined by CT Scan
Description: the primary outcome was evidence of existing tumor on pathologic review of the liver at the time or transplant or autopsy within the 18 month observational period. This outcome was compared to the CT HCC detection.
Time Frame: 18 months after start of therapy
Population: 14 cases (13 transplanted cases and 1 deceased case) had pathology available for review, representing 16 specimens (12 tumors in 14 livers))
Measure: Count of Units; unit: specimen
Units Other Than Participants: specimen
Groups:
- Tumor Free: No evidence of existing tumor was found on pathologic review of the liver at the time of transplant or autopsy within the 18 month observational period
- Tumor at Pathologic Review: Pathologic review found evidence of existing liver tumor at the time of transplant or autopsy within the 18 month observational period
Arm/Group | Tumor Free | Tumor at Pathologic Review
Number analyzed (Participants) | 4 | 10
Number analyzed (specimen) | 4 | 12
specimen
  CT negative (not seen) | 3 | 11
  CT Positive (seen) | 1 | 1
Statistical Analysis 1: Comparison: Tumor at Pathologic Review; Test type: Other; Sensitivity = 0.083, 95% CI 2-sided [0.00 to 0.38] — Twelve tumors were detected in the liver specimens, but only one of those was identified by the CT central readers
Statistical Analysis 2: Comparison: Tumor Free; Specificity; Test type: Other; Specificity = 0.75, 95% CI 2-sided [0.194 to 0.994] — The central CT readers correctly identified three out of the four patients without pathologic evidence of tumor

8. Secondary Outcome: Remote Tumor Occurrence Rates
Description: remote tumor occurrence rate is defined as a new intrahepatic tumor that developed remote from the ablation site within the 18 month period
Time Frame: 18 months after start of therapy
Measure: Number (95% Confidence Interval); unit: percent occuring
Arm/Group | Eligible Patients
Number analyzed (Participants) | 45
percent occuring | 0.53 [0.379 to 0.683]

9. Post Hoc Outcome: Rate of Successful Control of Disease at 18 Months, Including Transplants
Description: Outcome is positive (success) if the participant received a liver transplant or no diseaseis was observed by CT at 18 months after start of therapy Success rate it the fraction of eligible patients who are successes at 18 months.
Time Frame: 18 months after start of therapy
Measure: Number (95% Confidence Interval); unit: proportion of successes to eligible
Arm/Group | Eligible Patients
Number analyzed (Participants) | 45
proportion of successes to eligible | 0.51 [0.358 to 0.663]
Statistical Analysis 1: Comparison: Eligible Patients; Test type: Other — McNemar's Test to compare success rates after assuming transplants as successes versus after assuming transplants as failures; p = 0.0001, McNemar

ADVERSE EVENTS:
Time Frame: from initial ablation to 18 months
Groups:
- All Patients: patients with cirrhosis undergoing solitary or repetitive percutaneous RFA treatment sessions for the treatment of HCC.
  radiofrequency ablation
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 3/45
Serious Adverse Events (participants affected / at risk) | 5/45
Other Adverse Events (participants affected / at risk) | 26/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=45)
Death (Hepatobiliary disorders) | 2 (2) — Progression of disease
hemorrage with ablation/ procedure (Surgical and medical procedures) | 1 (1) — Post-Procedural hemorrage
Hematoma (Hepatobiliary disorders) | 1 (1) — Hematoma
Death (Hepatobiliary disorders) | 1 (1) — Multi organ failure
renal failure (Hepatobiliary disorders) | 1 (1) — Acute renal failure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=45)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1) — Bruising
Chills (General disorders) | 1 (1) — Chills
Hematoma (Blood and lymphatic system disorders) | 1 (1) — Hematoma
Hemorrhage with surgery (Blood and lymphatic system disorders) | 1 (1) — hemorrage with ablation/ procedure
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 3 (3) — Metabolic/Lab-Other LDH
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 1 (1) — Metabolic/Lab-Other AFP
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 2 (2) — Metabolic/Lab-Other ALT
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 1 (1) — Metabolic/Lab-Other ALT, SGPT
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 5 (5) — Metabolic/Lab-Other Ammonia
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 6 (7) — Metabolic/Lab-Other AST
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 1 (1) — Metabolic/Lab-Other AST,SGOT
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 4 (4) — Metabolic/Lab-Other Bilirubin
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 2 (2) — Metabolic/Lab-Other GGT
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 4 (4) — Metabolic/Lab-Other Hematocrit
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 3 (3) — Metabolic/Lab-Other Hemoglobin (Hgb)
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 1 (1) — Metabolic/Lab-Other HYPERGLYCEMIA
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 5 (6) — Metabolic/Lab-Other LDH
Pain (General disorders) | 2 (2) — Pain - Liver
Pain (General disorders) | 7 (9) — Pain - Other
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) — pneumothorax

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No